CLINICAL TRIAL: NCT07183774
Title: Does Sarcopenia Influence Rotator Cuff Tear Patterns? Radiological Insights From Patients With Rotator Cuff Syndrome
Status: Recruiting | Type: Observational
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sibel süzen Özbayrak, M.D, Haydarpasa Numune Training and Research Hospital
Other Study IDs: HNEAH-BAEK 2024/123
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tears; Sarcopenia; Shoulder Pain; Rotator Cuff Syndrome
Keywords: Rotator cuff syndrome; Rotator cuff tear; Sarcopenia
MeSH Terms: conditions — Rotator Cuff Injuries; Sarcopenia; Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with rotator cuff tear: Patients with parsiyel or full thickness rotator cuff tear in supraspinatus tendon
  Interventions: Diagnostic Test: Sarcopenia will be assessed using the STAR (Sonographic Thigh Adjustment Ratio) method.
- Patients without rotator cuff tear: Patients without tear in supraspnatus tendon
  Interventions: Diagnostic Test: Sarcopenia will be assessed using the STAR (Sonographic Thigh Adjustment Ratio) method.

INTERVENTIONS:
Diagnostic Test: Sarcopenia will be assessed using the STAR (Sonographic Thigh Adjustment Ratio) method. — A detailed evaluation of shoulder MRI scans will be conducted. The presence and severity of supraspinatus tendon tears, as well as the presence of muscle atrophy (assessed using the tangent sign), will be recorded. In addition, tears in other rotator cuff tendons, signs of tendinitis, and any other pathological findings will also be documented.
  Other Names: Shoulder MRIs of patients in each of these three categories will be analyzed to assess the presence, type, and severity of rotator cuff tears.

SUMMARY:
Sarcopenia is the loss of muscle mass due to aging, which consequently leads to a decline in muscle function. It is considered an independent risk factor for falls and fractures, disability, postoperative complications, and mortality. Rotator cuff tears are known to be influenced by systemic diseases such as diabetes, hypercholesterolemia, thyroid disorders, and osteoporosis. The aim of our study is to investigate whether there is a relationship between sarcopenia and rotator cuff tears, and if so, to determine the location and type of the tear.

DETAILED DESCRIPTION:
Patients aged between 40 and 75 years who present to the Physical Medicine and Rehabilitation Department's Shoulder Outpatient Clinic with shoulder pain lasting for at least three months, have undergone shoulder MRI as part of their diagnostic work-up, and have been clinically diagnosed with rotator cuff syndrome based on physical examination, will be included in the study.

Demographic data of the patients will be recorded. A detailed history regarding shoulder pain will be obtained. Pain severity will be assessed using the Visual Analog Scale (VAS), and shoulder functional impairment will be evaluated using the Shoulder Disability Questionnaire.

Following the clinical assessment of shoulder pain, sarcopenia evaluation will be performed by a different physician who is blinded to the patients' imaging and clinical findings. Sarcopenia will be assessed using the STAR (Sonographic Thigh Adjustment Ratio) method.

In this method, gait speed, handgrip strength (measured with a dynamometer), and the chair stand test will first be conducted. For gait speed, a 6-meter walking track will be used, and patients will be instructed to walk at their normal pace. The time will be recorded with a stopwatch, and each patient will perform the test three times, with the average recorded in meters per second (m/s).

In the chair stand test, the patient will be asked to rise from a chair five times as quickly as possible without using their arms, keeping both hands crossed over the chest (opposite shoulders). The time taken will be recorded with a stopwatch.

Handgrip strength will be measured using a Jamar dynamometer, with the shoulder in adduction, elbow at 90° flexion, and the wrist and hand in a neutral position. The patient will repeat the test three times, and the highest value will be recorded.

Patients will then be evaluated based on whether their gait speed is below 1.0 m/s, grip strength is 2 standard deviations below the norm, or chair stand time is ≥12 seconds.

Subsequently, anterior thigh muscle thickness will be measured using ultrasonography. Based on this comprehensive evaluation, patients will be categorized as non-sarcopenic, pre-sarcopenic, or sarcopenic.

At the end of the study, the shoulder MRIs of patients in each of these three categories will be analyzed to assess the presence, type, and severity of rotator cuff tears. This study aims to determine whether sarcopenia predisposes individuals to rotator cuff tears and, if so, what type of tear is more likely to occur in sarcopenic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with rotator cuff syndrome
2. Aged between 40 and 75 years

Exclusion Criteria:

1. History of previous shoulder surgery
2. Presence of shoulder pathology other than rotator cuff syndrome
3. History of surgical intervention involving the hip or thigh region
4. Being wheelchair-bound or bedridden
5. Presence of an oncologic disease
6. Diagnosis of any neurological disorder
7. Presence of cognitive impairment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study's target population will be patients aged 40 to 75 who have experienced shoulder pain for longer than three months and who have been physically evaluated and found to have rotator cuff syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
STAR value | Baseline
  Sarcopenia will be assessed using the STAR (Sonographic Thigh Adjustment Ratio) method.
  In this method, gait speed, handgrip strength (measured with a dynamometer), and the chair stand test will first be conducted. For gait speed, a 6-meter walking track will be used, and patients will be instructed to walk at their normal pace. The time will be recorded with a stopwatch, and each patient will perform the test three times, with the average recorded in meters per second (m/s).
  Subsequently, anterior thigh muscle thickness will be measured using ultrasonography. Based on this comprehensive evaluation, patients will be categorized as non-sarcopenic, pre-sarcopenic, or sarcopenic.

SECONDARY OUTCOMES:
Radiologic evaluation of shoulder MRI | Baseline
  Shoulder MRIs of patients in each of these three categories will be analyzed to assess the presence, type, and severity of rotator cuff tears.
  A detailed evaluation of shoulder MRI scans will be conducted. The presence and severity of supraspinatus tendon tears, as well as the presence of muscle atrophy (assessed using the tangent sign), will be recorded. In addition, tears in other rotator cuff tendons, signs of tendinitis, and any other pathological findings will also be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Haydarpaşa Numune Research and Training Hospital, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Atala NA, Bongiovanni SL, Galich AM, Bruchmann MG, Rossi LA, Tanoira I, Ranalletta M. Is sarcopenia a risk factor for rotator cuff tears? J Shoulder Elbow Surg. 2021 Aug;30(8):1851-1855. doi: 10.1016/j.jse.2020.10.001. Epub 2020 Nov 4. PMID 33157241
- [Result] Chung SW, Yoon JP, Oh KS, Kim HS, Kim YG, Lee HJ, Jeong WJ, Kim DH, Lee JS, Yoon JW. Rotator cuff tear and sarcopenia: are these related? J Shoulder Elbow Surg. 2016 Sep;25(9):e249-55. doi: 10.1016/j.jse.2016.02.008. Epub 2016 Apr 12. PMID 27083579
- [Result] Han DS, Wu WT, Hsu PC, Chang HC, Huang KC, Chang KV. Sarcopenia Is Associated With Increased Risks of Rotator Cuff Tendon Diseases Among Community-Dwelling Elders: A Cross-Sectional Quantitative Ultrasound Study. Front Med (Lausanne). 2021 May 5;8:630009. doi: 10.3389/fmed.2021.630009. eCollection 2021. PMID 34026779
- [Result] Kara M, Kara O, Durmus ME, Analay P, Sener FE, Citir BN, Korkmaz GO, Unlu Z, Tiftik T, Gurcay E, Mulkoglu C, Yalcinkaya B, Bagcier F, Aksakal MF, Erdogan K, Sertcelik A, Cakir B, Kaymak B, Ozcakar L. The Relationship Among Probable SARCopenia, Osteoporosis and SuprasPinatus Tendon Tears in Postmenopausal Women: The SARCOSP Study. Calcif Tissue Int. 2024 Apr;114(4):340-347. doi: 10.1007/s00223-024-01183-7. Epub 2024 Feb 12. PMID 38342790
- [Result] Kim JH, Jang I, Jeong S, Shin J, Yoon S, Lee H, Lee S. Examining the Relationship Between Sarcopenia and Rotator Cuff Tears: A Retrospective Comparative Study. J Clin Med. 2025 Jan 2;14(1):220. doi: 10.3390/jcm14010220. PMID 39797302